CLINICAL TRIAL: NCT05801666
Title: Acupuncture Effect on Dumping Syndrome in Esophagus Cancer Patients With Feeding Jejunostomy: A Study Protocol for A Single Blind Randomized Control Trial
Brief Title: Acupuncture Effect on Dumping Syndrome in Esophagus Cancer Patients With Feeding Jejunostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Peter Karl Mayer, Assistant Professor, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMU111-S-34
Record Dates: First submitted 2023-02-14; First posted 2023-04-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Esophagus Cancer; Acupuncture
Keywords: Esophagus Cancer; Acupuncture
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): Acupuncture points: ST36 (Zusanli), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Neiguan), and LI4 (Hegu) Liv 3(Taichung).
  Interventions: Other: Acupuncture
- Control group (Sham Comparator): Acupuncture on the sham points: ST36 (Zusanli), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Neiguan), and LI4 (Hegu) Liv 3(Taichung)(Sham 1~5). Those points are not indicated to treat digestion in Chinese medicine and in a location of 1 cm lateral/medial and 1 cm distal/proximal to those points there is no acupuncture point.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture 5 points

SUMMARY:
Esophagus cancer patients are at risk for malnourishment. Feeding jejunostomy is used in advanced esophagus cancer patients in order to support and supplement the patient's nutrition needs. In dumping syndrome, the food is rapidly introduced into the intestine at a rate that is faster than normal, it is associated with both digestive system and vasoactive symptoms. Dumping syndrome has an association with both esophagus cancer patients and feeding jejunostomy. In the mid and long term, dumping syndrome is an important issue that contributes to the risk of malnourishment in advanced esophagus cancer patients. Acupuncture effect on digestive symptoms was widely investigated with effective abilities to regulate and reduce digestive symptoms. Acupuncture is also considered a safe intervention for cancer patients.

A total of 60 advanced esophageal cancer patients will be divided into two equal groups, the intervention group (n=30) and the control groups (n=30). Patients in the Intervention group will receive acupuncture using the following acupoints: ST36 (Zusanli), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Neiguan), and LI4 (Hegu) liv 3 (Taichung). Patients and assessors will be blind to trial allocation. The patients in the Control group will receive shallow acupuncture on 12 non-acupoints (sham points). Both groups will receive acupuncture twice a week for 6 weeks. The main outcome measurements are body weight, BMI, the Sigstad's score and the Arts' dumping questionnaire, 3 and 6 months mortality.

DETAILED DESCRIPTION:
The direct effect of acupuncture on dumping syndrome was not previously well investigated. The goal of this randomized control clinical trial is to investigate the effect of acupuncture on dumping syndrome in esophagus cancer patients with jejunostomy tube feeding. We hypothesize that acupuncture will have a regulatory effect on dumping syndrome.

This research will investigate a possible cooperation and integration approach of both western and Chinese medicine in esophagus cancer treatment. In this integration, each treatment method focus on its strength (western medicine in tumor treatment and Chinese medicine in digestion symptoms) in order to improve the patient's condition and quality of life. This research will shed more light on the effectiveness of acupuncture as an intervention on both esophagus cancer patients and dumping syndrome. In case that the study findings will be in favor of acupuncture, it will provide a valuable, low cost supportive therapeutic option for advanced esophagus cancer patients with dumping syndrome.

This study will be conducted in the china medical university hospital in Taichung City, Taiwan, department of chest surgery. The study will be initiated after IRB approval and will be concluded until January 2024. Informed consent will be obtained prior to patient's enrollment. The 2 groups are an intervention group and a control group.

A total of 60 esophagus cancer patients with feeding jejunostomy from china medical hospital from the department of chest surgery. will be divided equally to 30 patients in each group after meeting the study inclusion criteria and informed consent.

60 patients from the china medical university will be divided into 2 groups. In both the ACU group and CON group, A qualified acupuncture doctor with at least 2 years of clinical experience will provide the intervention sessions on both groups. The acupuncture frequency will be 2 times a week for 6 weeks in both groups. Both groups will also receive routine western medicine treatments.

In addition to routine western medicine treatments, patients in the intervention group will also receive daily bilateral traditional Chinese medicine style acupuncture on the following acupuncture points: ST36 (Zusanli), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Neiguan), and LI4 (Hegu) liv 3(Taichung). The acupoints indications in this group are specific to treat indigestion-related conditions. The effectiveness of those points in treating digestion (with exception of liv 3(Taichung)) was shown in our previous research. The treatment will take place once a day, for 2 times a week for 6 weeks. A total of 12 needles will be used in each session. Acupuncture treatment will be performed with sterile needles manufactured by "Yu Kuang" acupuncture needles 40mm with 30G.

The patients in the control group will receive a bilateral shallow acupuncture (12 needles) on the sham points that are located 1 cm lateral/medial and 1 cm distal/proximal to the following acupoints: ST36 (Zusanli), ST37 (Shangjuxu), ST39 (Xiajuxu), PC6 (Neiguan), and LI4 (Hegu) liv 3 (Taichung) (figure 3). Those points are not indicated to treat digestion in Chinese medicine and in a location of 1 cm lateral/medial and 1 cm distal/proximal to those points there is no acupuncture point. The needle insertion will be a perpendicular shallow insertion into the skin tissue level. The acupuncture doctor will use the needle with tube insertion for needle insertion and will leave the needle in the depth of the tube insertion (approximately 4 mm depth into the skin) without needle manipulation. Needle retention time will be 30 minutes. In addition to the sham points, the patients in this group will also receive routine western medicine treatment as per each patient's needs. The treatment frequency and skin disinfection will be identical to the treatment group.

Main outcome measurements are: body weight, Body Mass Index (BMI) (will be measured weekly) dumping syndrome questioners: the Sigstad's score and the Arts' dumping questionnaire (will be measured on the baseline, week3, week 6).

The secondary outcomes are: muscle grip strength test (measured weekly) blood test: Complete Blood Count (CBC), kidney and electrolytes (measured as Adjuvant Concurrent Chemoradiation Therapy (CCRT) schedule), pre-albumin, albumin level, glucose blood levels, inflammation data including Erythrocyte Sedimentation Rate (ESR) and C-reactive Protein (CRP) (measured at baseline and on week 6).

Total Intensive care unit (ICU) stay, total hospital stay, total mechanical ventilation in days, will be measured 6 months after inclusion. Mortality will be measured at 3 months, 6 months. Medical charts and drug use will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Advanced esophageal cancer
* Post feeding jejunostomy
* Plan of CCRT for esophageal cancer

Exclusion Criteria:

* Acute infection
* Unstable vital signs
* Other medical conditions which would affect nutrition status

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Body Weight | baseline
  Unit: kg
Body Weight | week1
  Unit: kg
Body Weight | week2
  Unit: kg
Body Weight | week3
  Unit: kg
Body Weight | week4
  Unit: kg
Body Weight | week5
  Unit: kg
Body Weight | week6
  Unit: kg
Body Height | baseline
  Unit: cm
Body Height | week1
  Unit: cm
Body Height | week2
  Unit: cm
Body Height | week3
  Unit: cm
Body Height | week4
  Unit: cm
Body Height | week5
  Unit: cm
Body Height | week6
  Unit: cm
Body Mass Index | baseline
  BMI:kg/m*2
Body Mass Index | week1
  BMI:kg/m*2
Body Mass Index | week2
  BMI:kg/m*2
Body Mass Index | week3
  BMI:kg/m*2
Body Mass Index | week4
  BMI:kg/m*2
Body Mass Index | week5
  BMI:kg/m*2
Body Mass Index | week6
  BMI:kg/m*2
Sigstad's score | baseline
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week1
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week2
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week3
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week4
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week5
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Sigstad's score | week6
  Sigstad's score: diagnostic index >7 is suggestive of dumping syndrome. whereas a score <4 suggests that other diagnoses should be considered.(Shock +5, syncope/unconsciousness +4, Desire to lie or sit down +4, dyspnoea +3, Weakness/exhaustion +3, Sleepiness/drowsiness +3, Palpitation +3, Restlessness +2, Dizziness +2, Headaches +1, Feeling of warmth /sweating +1, Nausea +1, Abdominal fullness +1, Borborygmus +1, Eructation -1, Vomiting -4)
Arts' Dumping Questionnaire | baseline
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 1
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 2
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 3
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 4
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 5
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.
Arts' Dumping Questionnaire | week 6
  Each symptom is scored for severity on a 0-3 Likert scale (0=absent, 1=mild, 2=relevant and 3=severe), the total severity score for dumping syndrome is the sum of severities of all symptoms.

SECONDARY OUTCOMES:
Muscle grip strength test | baseline
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week1
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week2
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week3
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week4
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week5
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Muscle grip strength test | week6
  Electronic Hand Dyanmometer(EH101)), Unit: kg, Max Capacity: 90kg
Complete Blood Count (CBC)-WBC | baseline
  Unit:1000/μL
Complete Blood Count (CBC)-WBC | week 6
  Unit:1000/μL
Complete Blood Count (CBC)-RBC | baseline
  Unit:million/μL,
Complete Blood Count (CBC)-RBC | week 6
  Unit:million/μL,
Complete Blood Count (CBC)-Hemoglobin | baseline
  Unit:g/dL
Complete Blood Count (CBC)-Hemoglobin | week 6
  Unit:g/dL
Complete Blood Count (CBC)-Hematocrit | baseline
  Unit: %
Complete Blood Count (CBC)-Hematocrit | week 6
  Unit: %
Complete Blood Count (CBC)-MCV | baseline
  Unit: fL
Complete Blood Count (CBC)-MCV | week 6
  Unit: fL
Complete Blood Count (CBC)-MCH | baseline
  Unit: pg/cell
Complete Blood Count (CBC)-MCH | week 6
  Unit: pg/cell
Complete Blood Count (CBC)-MCHC | baseline
  Unit: g/dL
Complete Blood Count (CBC)-MCHC | week 6
  Unit: g/dL
Complete Blood Count (CBC)-RDW | baseline
  Unit: %
Complete Blood Count (CBC)-RDW | week 6
  Unit: %
Complete Blood Count (CBC)-Platelet | baseline
  Unit: 1000/μL
Complete Blood Count (CBC)-Platelet | week 6
  Unit: 1000/μL
Complete Blood Count (CBC)-PDW | baseline
  Unit: fL
Complete Blood Count (CBC)-PDW | week 6
  Unit: fL
Complete Blood Count (CBC)-MPV | baseline
  Unit: fL
Complete Blood Count (CBC)-MPV | week 6
  Unit: fL
Kidney and Electrolytes-eGFR | baseline
  Unit: mL/min/1.73m*2
Kidney and Electrolytes-eGFR | week 6
  Unit: mL/min/1.73m*2
Kidney and Electrolytes-Creatinine | baseline
  Unit: mg/dL
Kidney and Electrolytes-Creatinine | week 6
  Unit: mg/dL
Kidney and Electrolytes-ACR | baseline
  Unit: mg/g
Kidney and Electrolytes-ACR | week 6
  Unit: mg/g
Kidney and Electrolytes-Urea | baseline
  Unit: g/day
Kidney and Electrolytes-Urea | week 6
  Unit: g/day
Kidney and Electrolytes-Uric Acid | baseline
  Unit: mg/dL
Kidney and Electrolytes-Uric Acid | week 6
  Unit: mg/dL
Kidney and Electrolytes-Potassium | baseline
  Unit: mEq/L
Kidney and Electrolytes-Potassium | week 6
  Unit: mEq/L
Kidney and Electrolytes-Sodium | baseline
  Unit: mEq/L
Kidney and Electrolytes-Sodium | week 6
  Unit: mEq/L
Kidney and Electrolytes-Calcium | baseline
  Unit: mg/dL
Kidney and Electrolytes-Calcium | week 6
  Unit: mg/dL
Kidney and Electrolytes-Phosphate | baseline
  Unit: mg/dL
Kidney and Electrolytes-Phosphate | week 6
  Unit: mg/dL
Pre-Albumin | baseline
  Unit: mg/dL
Pre-Albumin | week 6
  Unit: mg/dL
Albumin level | baseline
  Unit: g/dL
Albumin level | week 6
  Unit: g/dL
Glucose blood levels | baseline
  Unit: mg/dL
Glucose blood levels | week 6
  Unit: mg/dL
Erythrocyte Sedimentation Rate (ESR) | baseline
  Unit: mm/h
Erythrocyte Sedimentation Rate (ESR) | week 6
  Unit: mm/h
C-reactive Protein (CRP) | baseline
  Unit: mg/L
C-reactive Protein (CRP) | week 6
  Unit: mg/L
Total Intensive care unit (ICU) stay, total hospital stay, total mechanical ventilation in days | measured at 6 months
  Hospital satistics
Mortality | measured at 3 months, 6 months
  Hospital statistics
Medical charts and drug use. | measured at 3 months, 6 months
  Hospital statistics

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mayer, Study Director — China Medical University,Taichung, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Mayer PK, Kao PY, Lee YC, Liao YF, Ho WC, Ben-Arie E. Acupuncture effect on dumping syndrome in esophagus cancer patients with feeding jejunostomy: A study protocol for a single blind randomized control trial. Medicine (Baltimore). 2023 Jun 9;102(23):e33895. doi: 10.1097/MD.0000000000033895. PMID 37335662